CLINICAL TRIAL: NCT00525928
Title: Assessment of Response to Open-label Treatment With Varenicline in Psychiatric Inpatients
Brief Title: Mood and Anti-craving Effects of Varenicline in Psychiatric Inpatients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficient recuirment
Sponsor: Butler Hospital (Other)
Collaborators: Brown University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0707-003
Record Dates: First submitted 2007-09-04; First posted 2007-09-06 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: Smoking; Depressive Disorder
Keywords: craving; smoking; depression
MeSH Terms: conditions — Smoking; Depressive Disorder; Depression | interventions — Varenicline

INTERVENTIONS:
Drug: varenicline — varenicline 0.5mg daily for days 1-3, 0.5mg twice daily for days 3-7, then 1mg twice daily for length of hospitalization
  Other Names: Chantix

SUMMARY:
This study of psychiatric inpatients will assess mood effects of varenicline, as well as assess if varenicline decreased nicotine cravings acutely.

This study will also measure side effects of varenicline when given in addition to other psychiatric and non-psychiatric medications.

DETAILED DESCRIPTION:
This study will measure mood effects and rapid anti-craving effects of varenicline in psychiatric inpatients. Patients will be offered to participate in the trial if they wish to stop smoking or wish to decrease nicotine cravings while in the hospital. They will not be able to use nicotine replacement products when taking varenicline.

Patients will be assessed with the QIDS-SR16, Minnesota Nicotine Withdrawal Scale as well as the Frequency, Intensity, and Burden of Side Effects (FISER) at baseline and daily during the trial; patients will be asked to enroll for the duration of their hospitalization. Patients will be assessed as to whether they wish to continue varenicline post-discharge.

ELIGIBILITY:
Inclusion Criteria:

1. Admission to Butler Hospital during study period.
2. Current tobacco users ages 18-65.
3. Able to give written, informed consent.

Exclusion Criteria:

1. Past adverse reaction to varenicline.
2. Treatment with varenicline on admission to Butler Hospital.
3. Renal failure or dialysis

(3) Current pregnancy or breastfeeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-10; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Estimated)

PRIMARY OUTCOMES:
improvement in Quick Inventory of Depressive Symptoms (QIDS-SR) | duration of hospitalization
improvement in Minnesota Nicotine Withdrawal Scale | days (duration of hospitalization)

SECONDARY OUTCOMES:
no significant intolerability, measured by the Frequency, Intensity, and Burden of Side Effects (FIBSER) and Adverse Events Checklist (SAFTEE-SI) | duration of hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Noah S Philip, MD, Principal Investigator — Butler Hospital; Lawrence H Price, MD, Study Director — Butler Hospital
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States